CLINICAL TRIAL: NCT03474848
Title: The Effects of Hand-Arm Bimanual Intensive Training (HABIT) in Hand Function and Daily Functioning of Children With Bilateral Cerebral Palsy: a Randomized Controlled Trial
Brief Title: The Effects of Hand-Arm Bimanual Intensive Training (HABIT) in Children With Bilateral Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, MARINA B BRANDAO, Professor, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HABIT_BilateralCP
Record Dates: First submitted 2018-03-15; First posted 2018-03-23 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; rehabilitation; hand function; daily functioning; hand-arm bimanual intensive training
MeSH Terms: conditions — Cerebral Palsy | interventions — Occupational Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HABIT (Experimental): Protocol of 90-hour of Hand-Arm Bimanual Intensive Training - 6 hours/day; 5 days/week, for 3 weeks
  Interventions: Other: HABIT
- Conventional Occupational Therapy (OT) (Active Comparator): Provision of 2 sessions/week (45 minutes), for 3 weeks
  Interventions: Other: Conventional Occupational Therapy (OT)

INTERVENTIONS:
Other: HABIT — Provision of individualized bimanual activities, individually chosen according to the child´s abilities, impairments and improvements in order to achieve success and to encourage bimanual use. Task difficulty is graded, focusing on enhancing the level of difficulty or speed, according to child's improvements. We use whole task practice (sequencing successive movements in the context of activities), part task practice (practice of specific components of the task in a repetitive sequence of time) and individualized functional goal training.
  Arms: HABIT
Other: Conventional Occupational Therapy (OT) — Children will maintain the occupational therapy sessions with their therapists, without any change in their routine at the rehabilitation center. Strategies such as functional training, stretching and sensory stimulation are used.
  Other Names: occupational therapy
  Arms: Conventional Occupational Therapy (OT)

SUMMARY:
Hand-Arm Bimanual Intensive Training (HABIT) has been shown to result in improvements in hand function and daily functioning of children with unilateral cerebral palsy (CP). Children with bilateral CP may also present difficulties to coordinate their hands to perform activities. Thus, HABIT may be a potential intervention for these individuals. We intend to examine the effects of HABIT on hand function and daily functioning of children with bilateral CP compared with conventional occupational therapy (OT). Our hypothesis is that children receiving HABIT will present larger improvements in manual dexterity and daily functioning as compared to conventional OT.

DETAILED DESCRIPTION:
Study Design: Randomized Controlled Trial. Study Participants & Setting: Forty children with bilateral CP recruited from the Associação Mineira de Reabilitação, Belo Horizonte, Brazil.

Procedures: After being included in the study, children will be randomly assigned to a intervention group (n=20) or a control group (n=20). Children in the intervention group will receive a 90-hour (6 hours/day; 5 days/week, 3 weeks) of Hand-Arm Bimanual Intensive Training (HABIT) while children in control group will maintain their usual frequency of Occupational Therapy (OT) sessions (45 minutes/session, twice a week, for 3 weeks), focusing on functional training, stretching and sensory stimulation. All participants will be assessed by an examiner blinded to group allocation before and after the intervention period, as well as 6 months after the intervention (follow-up).

Statistical Analysis: A 2 (groups) x 3 (assessments) analysis of variance will test the effects of group, assessment and group x assessment interaction with a level of significance set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Medical diagnosis of bilateral CP;
* Age between 4 and 17 years old;
* Manual Ability Classification System (MACS) ranging from levels I to III;
* Ability to understand verbal instructions.

Exclusion Criteria:

* Botulinum toxin or surgery in upper limbs in the previous 6 months of the study.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2016-01-05 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Functional goals | 6 months
  Canadian Occupational Performance Measure (COPM) - performance and satisfaction scales (each scale ranging 1-10; higher values, better outcomes)
Daily functioning | 6 months
  Pediatric Evaluation Disability Inventory (PEDI) [Scales: (1)self-care functional skills : ranging from 0-63; higher values, better outcomes; (2) caregiver assistance in self care: ranging from 0-40; higher values, better outcome]

SECONDARY OUTCOMES:
Manual dexterity | 6 months
  Jebsen Taylor Test of Hand Function (JTTHF): time to complete 6 hand function activities- score comprises the sum of time to complete the activities; ranging from 0-1080; higher values, worse outcome)
Bimanual hand use | 6 months
  Both Hand Assessment- score of bimanual hand function: score ranging from 0 to 100% (higher values, better outcome)
Manual dexterity | 6 months
  Box & Blocks Test (BBT)- number of blocks that are transported during 1 minute (there is no established max-min, higher values, better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Marina B Brandão, Doctor, Principal Investigator — Federal University of Minas Gerais

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Charles J, Gordon AM. Development of hand-arm bimanual intensive training (HABIT) for improving bimanual coordination in children with hemiplegic cerebral palsy. Dev Med Child Neurol. 2006 Nov;48(11):931-6. doi: 10.1017/S0012162206002039. PMID 17044964
- [Background] Gordon AM, Hung YC, Brandao M, Ferre CL, Kuo HC, Friel K, Petra E, Chinnan A, Charles JR. Bimanual training and constraint-induced movement therapy in children with hemiplegic cerebral palsy: a randomized trial. Neurorehabil Neural Repair. 2011 Oct;25(8):692-702. doi: 10.1177/1545968311402508. Epub 2011 Jun 23. PMID 21700924
- [Background] Bleyenheuft Y, Ebner-Karestinos D, Surana B, Paradis J, Sidiropoulos A, Renders A, Friel KM, Brandao M, Rameckers E, Gordon AM. Intensive upper- and lower-extremity training for children with bilateral cerebral palsy: a quasi-randomized trial. Dev Med Child Neurol. 2017 Jun;59(6):625-633. doi: 10.1111/dmcn.13379. Epub 2017 Jan 30. PMID 28133725
- [Background] Brandao MB, Ferre C, Kuo HC, Rameckers EA, Bleyenheuft Y, Hung YC, Friel K, Gordon AM. Comparison of Structured Skill and Unstructured Practice During Intensive Bimanual Training in Children With Unilateral Spastic Cerebral Palsy. Neurorehabil Neural Repair. 2014 Jun;28(5):452-61. doi: 10.1177/1545968313516871. Epub 2013 Dec 27. PMID 24376067
- [Background] de Brito Brandao M, Gordon AM, Mancini MC. Functional impact of constraint therapy and bimanual training in children with cerebral palsy: a randomized controlled trial. Am J Occup Ther. 2012 Nov-Dec;66(6):672-81. doi: 10.5014/ajot.2012.004622. PMID 23106987